CLINICAL TRIAL: NCT06252844
Title: The Impact of 6-months of Resistance Training on Intrinsic Capacity, Cognition, and Brain/Circulating Biomarkers of Neuroplasticity and Neuroinflammation in Older Adults With Mild Cognitive Impairment: a Randomized Controlled Trial.
Brief Title: The Impact of 6-months of Resistance Training on Brain and Muscle Health in Older Adults With MCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Collaborators: Lithuanian University of Health Sciences (Other); KU Leuven (Other); Vrije Universiteit Brussel (Other); Wingate Institute (Other); University of Hamburg-Eppendorf (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Vilma Dudoniene, Prof. Dr., Lithuanian Sports University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LithuanianSportsU-18
Record Dates: First submitted 2023-12-26; First posted 2024-02-12 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment; Older Adults at High Risk for MCI
Keywords: Mild Cognitive Impairment; Magnetic resonance imaging; Proton magnetic resonance spectroscopy (1H-MRS); Intrinsic capacity; Mobility; Blood biomarkers; cytokines; Neuroinflammation; Systemic inflammation; Neurometabolites
MeSH Terms: conditions — Cognitive Dysfunction; Neuroinflammatory Diseases | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Progressive resistance training (PRT) of lower limb muscles. Frequency of intervention: 2-3 times per week. Duration of intervention: 24 weeks.
  Interventions: Behavioral: Resistance exercise training
- Active control (Experimental): Flexibility training of the lower limb muscles. Frequency of intervention: 2-3 times per week. Duration of intervention: 24 weeks.
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: Resistance exercise training — Supervised PRT will consist of leg extension, leg curl, leg press, and calf raises. Initially participants will start with a 4 weeks adaptation with low loads at 15 (repetition maximum, RM) conducting for 1-3 sets. Further on subjects will continue with a 5 month of PRT with intensity increasing every 2 weeks from 12 to 6 RM. Each exercise will be done for 3 sets with 2 min rest periods between sets. After the 2 weeks at 6 RM, 1 week of rest will be applied. After the rest week, the same cycle starting from 12 RM will be repeated until the end of intervention.
  Arms: Intervention
Behavioral: Active control — Supervised static stretching exercises will be performed without causing an unpleasant feeling of stretching, up to pain, maintaining the stretching position for at least 30 s. Exercises will be performed slowly so that heart rate (HR) does not exceed 50% maximum. Subjects will calculate their HR before training, in the middle and after the training measuring the pulse for 10 s. Exercises will be repeated 3-5 times for each side of the body. The duration of the training will be match to PRT group and will take around 40 min. In order to keep the subjects interested and motivated, two of the stretching exercises will be changed every two weeks.
  Arms: Active control

SUMMARY:
The goal of this clinical trial is to learn about the effect of long resistance training intervention on brain and muscle health in older adults with mild cognitive impairment (MCI). The main question it aims to answer is whether progressive resistance training can prevent/delay neurodegenerative/pro-inflammatory processes that are detrimental to cognition, mobility, vitality, and mental health of older adults with MCI. Participants will undergo 6 months of supervise resistance training. Subjects in the intervention group will undergo sessions of structural and functional magnetic resonance imaging, proton magnetic resonance spectroscopy at baseline and end of intervention. Blood analyses and functional and cognitive tests will be performed at baseline after 3 months from the start of intervention and at the end of the intervention. Observations obtained from the intervention group will compare to data collected from age-matched active control group who will undergo flexibility training of lower limb muscles.

DETAILED DESCRIPTION:
Physical exercise appears to be effective in preventing transitions from normal cognitive aging to mild cognitive impairments (MCI) and from MCI to dementia-related disorders such as Alzheimer's disease (AD). The investigators will examine the longitudinal effects of progressive resistance training on biomarkers of (neuro)inflammation and neuroplasticity in a cohort of community-dwelling older individuals at high risk of developing MCI. The investigators will focus specifically on the effects of 24 weeks of resistance training on structural and neurochemical properties of the hippocampus and associations between exercise-induced changes in those properties and improvement in functional ability as quantified by pre-to-post changes in the mobility, cognition, psychological and vitality composites of intrinsic capacity (IC). Similarly, the investigators will examine the association between exercise-induced changes in global internal capacity index and exercise-induced changes in the expressions of inflammatory biomarkers (specifically, IL-1β, IL-6, IL-10, IL-18, kynurenine, and TNFa), myokines (specifically, BDNF, IGF-1, irisin), and circulating biomarkers of neurodegeneration (specifically, neurofilament light chain - NfL), tauopathy (specifically, total and phosphorylated tau181) and amyloid pathology (specifically, Aβ42/Aβ40 ratio). Blood samples will be collected between 8 a.m. and 11 a.m. after fasting. Behavioral outcome measures from gait/balance tests, handgrip strength test, cognitive tests, psychological tests, etc. and serum/plasma levels of the circulating biomarkers will be assessed at baseline, mid-intervention time (12 weeks), immediately post-intervention time (24 weeks), and at six-month follow-up (48 weeks). Structural MRI (sMRI) images, diffusion MRI (dMRI) images, resting state functional MRI (rs-fMRI) data and proton magnetic resonance spectroscopy (1H-MRS) data from the brain and T1-wighted images and 1H-MRS spectra from the lower-limb musculature will be collected at baseline and immediately post-treatment time (24 weeks) using a Siemens 3T Skyra scanner. Findings from this study will be used to provide evidence-based frameworks for implementation of longitudinal exercise interventions in prevention of dementia-related neurodegenerative disease among older with MCI. Further, the investigators will assess the effects of exercise on longitudinal changes in muscle mass, muscle strength, and neuromuscular functioning and examine the associations between these changes and exercise induced changes in locomotion capacity and postural stability as well as the prevention of sarcopenia and frailty. Secondary (exploratory) outcome measures will be (1) effects of the longitudinal strength training program on brain structural and neurochemical properties and (2) demographic factors, physiological properties and/or biomarkers that predict response to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 65+ years old,
* Community-dwelling,
* Sedentary (not engaged in any structured activity for exercise) or non-sedentary individuals who engaged in mild recreational activities for less than 150 min/week.
* A score of 18 to 25 on the Montreal Cognitive Assessment (MoCA) with or without a diagnosis of MCI. The diagnosis of MCI will be confirmed by a qualified mental health care specialist at the screening evaluation according to the International Classification of Diseases (ICD-10) and the Petersen criteria (Petersen et al, 2014).
* Fluent in Lithuanian.

Exclusion Criteria:

* Age < 65 years.
* MoCA ≥ 26 or MoCA < 18,
* Symptomatic heart or cardiopulmonary disorders, diabetes, diagnosis of renal/hepatic disease, oncology, brain injury, diagnosis of neurologic, psychiatric, or musculoskeletal diseases.
* Physical or orthopedic conditions (rheumatic symptoms, chronic pain, fractures, acute muscle injuries) that limit the subject's ability to participate in the training program.
* Moderate to severe intake of alcohol (intake of 3 drinks or more/day for men and 2 drink or more/day for women).
* Current smoker
* Intake of drugs or psychiatric medications.
* Contraindications to perform MRI (e.g., claustrophobia, cardiac pacemaker, internal pacing wires, metal implants, etc.).
* Body mass index (BMI) > 35 kg/m2 or body weight > 130 kg.
* Participation in routine exercise or physical activities (IPAQ).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in intrinsic capacity | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Assessment of intrinsic capacity subdomains will be conducted according to the WHO ICOPE guidelines.
  Outcome measures:
  Locomotion capacity [scale 0 to 12] with higher scores indicating a better outcome.
  Cognition capacity [scale: 0 to 4], with higher scores indicating a better outcome.
  Psychological capacity (mood) [scale: 0 to 4] with higher scores indicating a better outcome.
  Vitality [scale 0 to 12], with higher scores indicating a better outcome. Sensory capacity index [scale 0 to 3], with higher scores indicating a better outcome.
  Capacity indexes for each of the above mentioned subdomains will be calculated as the scores obtained divided by the maximum possible scores [scale 0 to 1].
  The global intrinsic capacity index will be calculated as the sum of the subdomain's capacity indexes [scale 0 to 5] with higher scores indicating a better outcome.
Changes in global cognition | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Outcome measure: scores on the Montreal cognitive assessment (MoCA) [range 0 - 30] with higher scores indicating better performance.
Changes in psychological assessment of depression | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Outcome measure: scores on the Geriatric depression scale (GDS), [range 0-15] with higher score indicate severe depression.
Changes in reaction time | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  ANAM4 cognitive test battery, including:
  Go/No-Go test (GNG), 6 Letter Memory Search test (6LMST), Manikin test (MNKT)
  Outcome measures: Reaction Time (in milliseconds) with shorter time indicating a better outcome.
Changes in reaction accuracy | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  ANAM4 cognitive test battery, including:
  Go/No-Go test (GNG), 6 Letter Memory Search test (6LMST), Manikin test (MNKT)
  Outcome measures: % number of correct responses with higher value indicating a better outcome.
Changes in cognitive efficiency | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  ANAM4 cognitive test battery, including:
  Go/No-Go test (GNG), 6 Letter Memory Search test (6LMST), Manikin test (MNKT)
  Outcome measures: throughput (= number of correct responses divided by mean RT for correct responses) with higher value indicating a better outcome
Changes in Stroop interference score | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Stroop Color and Word test (SCWT)
  Outcome measure:
  interference score (in seconds) Interference = CWT - [(WT + CT)/2] where WT, CT, and CWT are times (in seconds) to complete the Word, Color, and Color-Word conditions, respectively. Lower interference score indicates a better outcome.
Changes in performance on the Trail Making Test (TMT) | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Complete parts A and part B of the Trail Making Test
  Outcome measures:
  Time (in seconds) required to complete part A (Trail A scores) Time (in seconds) required to complete part B (Trail B scores) Shorter time indicated a better outcome.
Changes in sway velocity | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Center of pressure (CoP) data will be collected in stance position with a single piezoelectric force plate (KISTLER, model 9286) under single and dual-task condition.
  Outcome measures:
  CoP sway velocity (CoPv) in ML and AP sway directions (millimiter/seconds). Lower sway velocity represents a better outcome.
Changes in dual-task cost for sway velocity | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Dual task cost (DTC) will be quantified as % change of sway velocity from dual to single task relative to their single task values.
  Increased negative value represents a better outcome whereas increased positive value represents a worse outcome.
Changes in agility | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  8-Foot timed up and go (8-foot TUG): Outcome measure: time to complete the task in seconds. Shorter time to complete the task represents a better outcome.
Changes in lower body strength and muscular endurance | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  30s Chair-Rise test: Outcome measure: number of sit-to-stand repetitions completed in 30 seconds. More sit-to-stand repetitions represents a better outcome.
Changes in levels of Albumin (Alb) | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Albumin levels [grams/deciliter (g/dL)] will be measured with GBC-system XN-1500 blood analyzer. Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional.
Changes in levels of Hemoglobin (Hb) | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Hemoglobin levels [grams/deciliter (g/dL)] will be measured with GBC-system XN-1500 blood analyzer. Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional.
Changes in levels of C-reactive protein (CRP) | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  CRP levels [milligrams/deciliter (mg/dL)] will be measured with COBAS PRO blood analyzer. Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional.
Changes in circulating levels of cytokines | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Serum levels of the interleukins IL-1β, IL-6, IL-10, IL-18 and serum levels of TNFα [all picograms/milliliter(pg/ml)] will be assessed with enzyme-linked immunosorbent assay (ELISA). Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional. Serum samples will be stored in the refrigerator compartment of the laboratory of the Lithuanian Sports University at -80 degrees Celsius until further analysis.
Changes in circulating levels of Kynurenine | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Serum levels of Kynurenine [nanograms/milliliter(ng/ml)] will be assessed with enzyme-linked immunosorbent assay (ELISA). Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional. Serum samples will be stored in the refrigerator compartment of the laboratory of the Lithuanian Sports University at -80 degrees Celsius until further analysis.
Changes in circulating levels of brain-derived neurotrophic factor (BDNF) | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Plasma levels of BDNF [picograms/milliliter(pg/mL)] will be assessed with enzyme-linked immunosorbent assay (ELISA). Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional. Plasma samples will be stored in the refrigerator compartment of the laboratory of the Lithuanian Sports University at -80 degrees Celsius until further analysis.
Changes in circulating levels of Insulin-like growth factor 1 (IGF-1) | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Serum levels of IGF-1 [nanograms/milliliter(pg/mL)] will be assessed with enzyme-linked immunosorbent assay (ELISA). Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional. Serum samples will be stored in the refrigerator compartment of the laboratory of the Lithuanian Sports University at -80 degrees Celsius until further analysis.
Changes in circulating levels of Irisin | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Plasma levels of irisin [nanograms/milliliter (ng/ml)] will be assessed using enzyme-linked immunosorbent assay (ELISA). Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional. Serum samples will be stored in the refrigerator compartment of the laboratory of the Lithuanian Sports University at -80 degrees Celsius until further analysis.
Changes in circulating levels of c-terminal agrin fragment-22 (CAF22) | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Serum levels of c-terminal agrin fragment-22 [picograms/milliliter (pg/ml)] will be assessed using enzyme-linked immunosorbent assay (ELISA). Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional. Serum samples will be stored in the refrigerator compartment of the laboratory of the Lithuanian Sports University at -80 degrees Celsius until further analysis.
Changes in circulating levels of Neurofilament light chain (NfL) | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Plasma levels of NfL (picograms/milliliter (pg/ml)] will be assessed using enzyme-linked immunosorbent assay (ELISA). Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional. Plasma samples will be stored in the refrigerator compartment of the laboratory of the Lithuanian Sports University at -80 degrees Celsius until further analysis.
Changes in circulating levels of tau proteins | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Plasma levels of phosphorylated tau181 (p-tau181) and total tau (t-tau) [both, picograms/milliliter (pg/ml)] will be assessed using enzyme-linked immunosorbent assay (ELISA). Blood samples will be collected at the at antecubital vein after 12-h fasting by a qualified medical professional. Plasma samples will be stored in the refrigerator compartment of the laboratory of the Lithuanian Sports University at -80 degrees Celsius until further analysis.
Changes in circulating levels of beta amyloids | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Plasma levels of beta amyloid 40 (Aβ40) and beta amyloid 42 (Aβ42) will be assessed using enzyme-linked immunosorbent assay (ELISA). Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional. Plasma samples will be stored in the refrigerator compartment of the laboratory of the Lithuanian Sports University at -80 degrees Celsius until further analysis. Plasma levels of Aβ40 and Aβ42 will be combined to calculate the Aβ42/40 ratio.
Changes in brain volume properties | Baseline and Post-intervention time (24 weeks); Optional: follow-up at 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Whole brain T1-weighted images, T2-wighted images, T2* relaxation images and fluid attenuated inversion recovery (FLAIR) images will be obtained. Outcome measures will be grey matter (GM) volumes, white matter (WM) volumes (WM) and WM hyperintensity (WMH) volumes [all in cubic millimeter (mm^3)] of cortical and subcortical structures. A total WMH volume will be obtained by summing the volumes of hyperintensities from all of the substructures. A large WMH volume will be taken as an indicator for cerebrovascular abnormalities. Image processing: FreeSurfaer software, version 6 (freely available).
Changes in brain cortical thickness | Baseline and Post-intervention time (24 weeks); Optional: follow-up at 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Whole brain T1-weighted images. Outcome measures: GM cortical thicknesses (in mm) of cortical substructures. Image processing: FreeSurfer software, version 6 (freely available).
Changes in brain WM microstructural organization | Baseline and Post-intervention time (24 weeks); Optional: follow-up at 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Participants will undergo whole brain diffusion-weighted imaging (DWI). Outcome measures will be the Fractional anisotropy (FA) of WM tracts in the brain. Image processing will be possible with the use of the ExploreDTI software (freely available).
Changes in brain neurometabolic levels | Baseline and Post-intervention time (24 weeks); Optional: follow-up at 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Single voxel proton magnetic resonance spectroscopy (1H-MRS) of left hippocampus (HPC), right dorsolateral prefrontal cortex (dlPFC) and left sensory motor cortex (SM1). Data will be processed with LC Model within the Osprey pipeline (freely available).
  Outcome measures will be the water-referenced levels of:
  * N-acetyl aspartate (NAA),
  * Creatine (Cr),
  * Choline (Cho),
  * Myoinositol (mIns),
  * Glutamine-glutamate complex (Glx),
  All levels are expressed in institutional units (i.u).
Changes in brain neurometabolic ratios | Baseline and Post-intervention time (24 weeks); Optional: follow-up at 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Single voxel proton magnetic resonance spectroscopy (1H-MRS). Ratios will be calculated from water-referenced levels of NAA, Cho, mIns, Glx, and Cr in left Hippocampus, left sensorimotor cortex and right dorsolateral prefrontal cortex.
  Outcome measures:
  * NAA/Cr,
  * Cho/Cr,
  * mIns/Cr,
  * Glx/Cr
  * NAA/mIns
  Ratios are expressed in arbitrary units (a.u).
Changes in quadriceps/hamstrings cross sectional area | Baseline and Post-intervention time (24 weeks); Optional: follow-up at 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  T1-weighted images of the left/right thighs
  Outcome measures:
  * Quadricepscross-sectional areas at mid-thigh (in cm^2)
  * Hamstring cross-sectional areas at mid-thigh (in cm^2).
Changes in quadriceps myocellular lipid content | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  1H-MRS spectra from the right quadriceps.
  Outcome measures:
  * Quadriceps intramyocellular lipid (IMCL) content (% of unsuppressed water signal area)
  * Quadriceps extramyocellular lipid (EMCL) content (% of unsuppressed water signal area).
  * Quadriceps total IMCL and EMCL content (% of unsuppressed water signal area)
Changes in body composition and BMI | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  TANITA body impedance analysis. Outcome measures: total body weight, body fat mass, lean muscle mass, and bone mass (in kilograms).
  Total body weight and fat weight will be combined to calculate % body fat. Total body weight and height will be combined to calculate the body mass index (BMI) in kilograms/meter^2.
Changes in knee muscle torque production | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Biodex
  * Maximum voluntary contraction (MVC) torque during isometric contraction in Newton/meter (N/m).,
  * Knee extension/flexion concentric isokinetic peak torques (PT) in N/m at isokinetic speed of 60 and 180 deg/s.
  * Torque development in N/m at 30ms, 50 ms, 100 ms, and 200 ms from onset of contraction.
Changes in muscle contraction time | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Tensiomyography (TMG) of left and right rectus femoris (RF) and biceps femoris (BF) heads.
  Outcome measures:
  Delay time (Td) and contraction time (Tc) of left/right RF and BF (in milliseconds).
Changes in muscle contraction displacement | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Tensiomyography (TMG) of left and right rectus femoris (RF) and biceps femoris (BF) heads.
  Outcome measures:
  Muscle contraction displacement (Dm) of left/right RF and BF (in millimeter).
Changes in muscle contraction velocity | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Tensiomyography (TMG) of left and right rectus femoris (RF) and biceps femoris (BF) heads.
  Muscle contraction displacement (Dm), delay time (Td) and contraction time (Tc) will be combined to calculate contraction velocity (Vc) of left/right RF and BF.
  Vc = [Dm/(Td +Tc)] (in millimeter/second).
Changes in level of fatigue | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Participants will complete the Multidimensional Fatigue Inventory (MFI-20) [range 4-20] with higher scores indicate a higher level of fatigue.
Changes in level of frailty | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Subjects will undergo the Edmonton Frail Scale survey [range 0 -17] with higher scores indicate a higher level of frailty.
Changes in health status | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Participants will complete the 36-Items Form Health survey (SF-36), [range 0-100] with higher score indicate better physical and mental health.
Changes in nutritional status | Baseline, Mid-intervention time (12 weeks) and Post-intervention time (24 weeks); Optional: follow-up at 48 weeks (1st follow-up) and 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Participants will complete the Mini Nutritional Assessment (MNA) survey [range 0-14] with higher score indicate better nutritional condition.

SECONDARY OUTCOMES:
Changes in blood count | Baseline and Post-intervention time (24 weeks); Optional follow-up at 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Blood count tests will be conducted using GBC-system XN-1500 blood analyzer. Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional.
  Outcome measures:
  * Red blood cell count measured in cells per liter (cells/L). Normal range [Male: 4.35 x 10^12 to 5.65 x 10^12 cells/L; Female: 3.92 x 10^12 to 5.13 x 10^12 cells/L].
  * White blood cell count measured in cells per liter (cells/L). Normal range [3.4 x 10^9 to 9.6 x 10^9 cells/L].
  * Platelet count measured in cells per liter (cells/L). Normal range [Male: 135 x 10^9 to 317 10^9 cells/L; Female: 157 x 10^9 to 371x10^9 cells/L].
  * Hematocrit (percentage by volume of red cells). Normal range [Male: 38.3% to 48.6%; Female: 35.5% to 44.9%].
Changes in lipid profiles | Baseline and Post-intervention time (24 weeks); Optional follow-up at 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  A lipidogram test will be conducted using COBAS PRO blood analyzer. Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional.
  Outcome measures:
  * Level of HDL (high-density lipoprotein) cholesterol [millimole/liter (mmol/L)]. Normal range < 1.68 mmol/L
  * Level of LDL (high-density lipoprotein) cholesterol. Normal range < 2.59 mmol/L.
  * Level of total cholesterol. Normal range < 5.2 mmol/L
  * Level of Triglycerides. Normal range < 1.7 mmol/L
Changes in Glycosylated Hemoglobin (HbA1c) | Baseline and Post-intervention time (24 weeks); Optional follow-up at 72 weeks (2nd follow-up) for participants who would be willing to continue their training.
  Glycosylated Hemoglobin levels will be measured using the Alinity C method. Blood samples will be collected at the antecubital vein after 12-h fasting by a qualified medical professional.
  Outcome measures:
  - Level of HbA1c [millimole/liter (mmol/L)]. Normal range < 42 mmol/L (~ 6%).
Self-report measure of habitual physical activity | Baseline
  Participants will complete the International Physical Activity Questionnaire (IPAQ-LT). Higher score indicate high physical activity level.

CONTACTS AND LOCATIONS:
Overall Officials: Oron Levin, PhD, Principal Investigator — Lithuanian Sports University
Locations (2):
- Lithuania (2):
  - Institute of Sport Science and Innovations, Kaunas
  - Lithuanian Sports University, Kaunas

IPD SHARING:
Plan to Share IPD: Yes
1. The data collected in this study will be available to all collaborators in an interactive closed data repository.
  2. Analyzed data will be available in an open-source data repository for all researchers upon request after the end of the study.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data sharing with collaborators: at the end of data collection (anticipated: February 2025) Data sharing with other researchers: one months after publication (anticipated: June 2026)
Access Criteria: Data collected and additional supporting information will be shared unconditionally with all collaborators upon signing a Data Sharing Agreement.
  Access to the open-source data repository will be granted by the principal investigator and/or study manager.

REFERENCES:
- [Background] Bautmans I, Knoop V, Amuthavalli Thiyagarajan J, Maier AB, Beard JR, Freiberger E, Belsky D, Aubertin-Leheudre M, Mikton C, Cesari M, Sumi Y, Diaz T, Banerjee A; WHO Working Group on Vitality Capacity. WHO working definition of vitality capacity for healthy longevity monitoring. Lancet Healthy Longev. 2022 Nov;3(11):e789-e796. doi: 10.1016/S2666-7568(22)00200-8. PMID 36356628
- [Background] Beard JR, Si Y, Liu Z, Chenoweth L, Hanewald K. Intrinsic Capacity: Validation of a New WHO Concept for Healthy Aging in a Longitudinal Chinese Study. J Gerontol A Biol Sci Med Sci. 2022 Jan 7;77(1):94-100. doi: 10.1093/gerona/glab226. PMID 34343305
- [Background] Belloni G, Cesari M. Frailty and Intrinsic Capacity: Two Distinct but Related Constructs. Front Med (Lausanne). 2019 Jun 18;6:133. doi: 10.3389/fmed.2019.00133. eCollection 2019. PMID 31275941
- [Background] Cesari M, Araujo de Carvalho I, Amuthavalli Thiyagarajan J, Cooper C, Martin FC, Reginster JY, Vellas B, Beard JR. Evidence for the Domains Supporting the Construct of Intrinsic Capacity. J Gerontol A Biol Sci Med Sci. 2018 Nov 10;73(12):1653-1660. doi: 10.1093/gerona/gly011. PMID 29408961
- [Background] Cesari M, Sadana R, Sumi Y, Amuthavalli Thiyagarajan J, Banerjee A. What Is Intrinsic Capacity and Why Should Nutrition Be Included in the Vitality Domain? J Gerontol A Biol Sci Med Sci. 2022 Jan 7;77(1):91-93. doi: 10.1093/gerona/glab318. No abstract available. PMID 35015816
- [Background] De Luca A, Kuijf H, Exalto L, Thiebaut de Schotten M, Biessels GJ; Utrecht VCI Study Group. Multimodal tract-based MRI metrics outperform whole brain markers in determining cognitive impact of small vessel disease-related brain injury. Brain Struct Funct. 2022 Sep;227(7):2553-2567. doi: 10.1007/s00429-022-02546-2. Epub 2022 Aug 22. PMID 35994115
- [Background] Gallardo-Gomez D, Del Pozo-Cruz J, Noetel M, Alvarez-Barbosa F, Alfonso-Rosa RM, Del Pozo Cruz B. Optimal dose and type of exercise to improve cognitive function in older adults: A systematic review and bayesian model-based network meta-analysis of RCTs. Ageing Res Rev. 2022 Apr;76:101591. doi: 10.1016/j.arr.2022.101591. Epub 2022 Feb 17. PMID 35182742
- [Background] Leung AYM, Su JJ, Lee ESH, Fung JTS, Molassiotis A. Intrinsic capacity of older people in the community using WHO Integrated Care for Older People (ICOPE) framework: a cross-sectional study. BMC Geriatr. 2022 Apr 8;22(1):304. doi: 10.1186/s12877-022-02980-1. PMID 35395736
- [Background] Levin O, Netz Y, Ziv G. The beneficial effects of different types of exercise interventions on motor and cognitive functions in older age: a systematic review. Eur Rev Aging Phys Act. 2017 Dec 21;14:20. doi: 10.1186/s11556-017-0189-z. eCollection 2017. PMID 29276545
- [Background] Levin O, Vints WAJ, Ziv G, Katkute G, Kusleikiene S, Valatkeviciene K, Sheoran S, Drozdova-Statkeviciene M, Gleizniene R, Paasuke M, Dudoniene V, Himmelreich U, Cesnaitiene VJ, Masiulis N. Neurometabolic correlates of posturography in normal aging and older adults with mild cognitive impairment: Evidence from a 1H-MRS study. Neuroimage Clin. 2023;37:103304. doi: 10.1016/j.nicl.2022.103304. Epub 2022 Dec 24. PMID 36580713
- [Background] Netz Y. Is There a Preferred Mode of Exercise for Cognition Enhancement in Older Age?-A Narrative Review. Front Med (Lausanne). 2019 Mar 29;6:57. doi: 10.3389/fmed.2019.00057. eCollection 2019. PMID 30984760
- [Background] Petersen RC, Caracciolo B, Brayne C, Gauthier S, Jelic V, Fratiglioni L. Mild cognitive impairment: a concept in evolution. J Intern Med. 2014 Mar;275(3):214-28. doi: 10.1111/joim.12190. PMID 24605806
- [Background] Sheoran S, Vints WAJ, Valatkeviciene K, Kusleikiene S, Gleizniene R, Cesnaitiene VJ, Himmelreich U, Levin O, Masiulis N. Strength gains after 12 weeks of resistance training correlate with neurochemical markers of brain health in older adults: a randomized control 1H-MRS study. Geroscience. 2023 Jun;45(3):1837-1855. doi: 10.1007/s11357-023-00732-6. Epub 2023 Jan 26. PMID 36701005
- [Background] Tatebe H, Kasai T, Ohmichi T, Kishi Y, Kakeya T, Waragai M, Kondo M, Allsop D, Tokuda T. Quantification of plasma phosphorylated tau to use as a biomarker for brain Alzheimer pathology: pilot case-control studies including patients with Alzheimer's disease and down syndrome. Mol Neurodegener. 2017 Sep 4;12(1):63. doi: 10.1186/s13024-017-0206-8. PMID 28866979
- [Background] Vints WAJ, Gokce E, Langeard A, Pavlova I, Cevik OS, Ziaaldini MM, Todri J, Lena O, Sakkas GK, Jak S, Zorba Zormpa I, Karatzaferi C, Levin O, Masiulis N, Netz Y. Myokines as mediators of exercise-induced cognitive changes in older adults: protocol for a comprehensive living systematic review and meta-analysis. Front Aging Neurosci. 2023 Jul 13;15:1213057. doi: 10.3389/fnagi.2023.1213057. eCollection 2023. PMID 37520128
- [Background] Vints WAJ, Levin O, Fujiyama H, Verbunt J, Masiulis N. Exerkines and long-term synaptic potentiation: Mechanisms of exercise-induced neuroplasticity. Front Neuroendocrinol. 2022 Jul;66:100993. doi: 10.1016/j.yfrne.2022.100993. Epub 2022 Mar 11. PMID 35283168
- [Background] Vints WAJ, Kusleikiene S, Sheoran S, Sarkinaite M, Valatkeviciene K, Gleizniene R, Kvedaras M, Pukenas K, Himmelreich U, Cesnaitiene VJ, Levin O, Verbunt J, Masiulis N. Inflammatory Blood Biomarker Kynurenine Is Linked With Elevated Neuroinflammation and Neurodegeneration in Older Adults: Evidence From Two 1H-MRS Post-Processing Analysis Methods. Front Psychiatry. 2022 Apr 11;13:859772. doi: 10.3389/fpsyt.2022.859772. eCollection 2022. PMID 35479493
- [Background] Kothapalli SVVN, Benzinger TL, Aschenbrenner AJ, Perrin RJ, Hildebolt CF, Goyal MS, Fagan AM, Raichle ME, Morris JC, Yablonskiy DA. Quantitative Gradient Echo MRI Identifies Dark Matter as a New Imaging Biomarker of Neurodegeneration that Precedes Tisssue Atrophy in Early Alzheimer's Disease. J Alzheimers Dis. 2022;85(2):905-924. doi: 10.3233/JAD-210503. PMID 34897083
- See also: Guidance on person-centred assessment and pathways in primary care — https://apps.who.int/iris/bitstream/handle/10665/326843/WHOFWC-ALC-19.1-eng.pdf?sequence=17&isAllowed=y
- See also: Resistance Training for Older Adults: Position Statement From the National Strength and Conditioning Association — https://doi.org/10.1519/jsc.0000000000003230